CLINICAL TRIAL: NCT05095389
Title: Adipose Derived Regenerative Cells (ADRCs) in the Treatment of Diabetic Foot Ulcers: a Prospective, Double-blind, Multi-center, Randomized, Parallel-group Study
Brief Title: Adipose Derived Regenerative Cells In the Treatment of Diabetic Foot Ulcers
Acronym: ASCEND
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Paracrine, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-01
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; DFU; Non-healing Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel-Group, Double-Blind, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo is visually indistinguishable from Active Treatment. Every patient receives Standard Care, plus either Active Treatment or Placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Standard Care plus ARDCs (Experimental): * All patients will undergo small volume liposuction, and adipose tissue harvested will be processed to ADRCs during same procedure.
  * All patients will receive standard care for their Diabetic Foot Ulcer.
  * Additionally, patients randomized to the ADRC arm will receive ADRCs
  Interventions: Device: ADRCs; Other: standard care
- Standard Care plus Placebo (Active Comparator): * All patients will undergo small volume liposuction, and adipose tissue harvested will be processed to ADRCs during same procedure.
  * All patients will receive standard care for their Diabetic Foot Ulcer.
  * Additionally, patients randomized to the Control arm will receive Placebo
  Interventions: Other: standard care; Other: Placebo

INTERVENTIONS:
Device: ADRCs — Administration of Autologous Adipose Derived Regenerative Cells into the Diabetic Foot Ulcer
  Arms: Standard Care plus ARDCs
Other: standard care — standard care
Other: Placebo — placebo
  Arms: Standard Care plus Placebo

SUMMARY:
A Prospective, Double-blind, Multi-center, Randomized, Parallel-group safety and efficacy study of adipose-derived regenerative cells (ADRCs) in the treatment of patients with diabetic foot ulcers (DFU).

DETAILED DESCRIPTION:
Subjects will have at least one diabetic foot ulcer between 1 cm2 and 16 cm2 area that remains open despite at least 30 days of DFU care and will need debridement as a part of their care.

Subjects will be randomly assigned to one of two groups (ADRC Group will receive standard care plus ADRC, and Control Group will receive standard care plus matched placebo).

ADRCs will be harvested from a small volume liposuction performed on the same day as, but prior to, the debridement procedure. Fat harvest will occur through small volume (approximately 100-200 mL) liposuction prior to the surgical debridement procedure on the same day as the planned autograft procedure.

The lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs for application to an autograft site. Cells will be delivered via direct injection (minimal wound penetration with a 22 gauge needle, total volume 5 mL) into the DFU (injected around the circumference and applied to the base of the ulcer).

ELIGIBILITY:
Inclusion Criteria:

* T1D or T2D
* Diabetic Foot Ulcer, from 1 to 12 months in duration
* Wagner Grade 1 or Superficial 2
* Adequate perfusion
* Able to undergo liposuction

Exclusion Criteria:

* Diabetic Foot Ulcer penetrates to capsule, tendon, or bone
* Active infection
* Non-diabetic neuropathy
* Significant cardiovascular event within 6 months before screening

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
DFU Closure Rate | 12 Weeks
  The rate of closure at 12 Weeks

SECONDARY OUTCOMES:
Percent Reduction of Wound Area | 12 Weeks
  Percent Reduction of Wound Area from Baseline to 12 Weeks for Ulcers not Completely Healed

IPD SHARING:
Plan to Share IPD: No
No IPD/PHI will be made available